CLINICAL TRIAL: NCT05145335
Title: Perceptual, Hemodynamic and Cardiovascular Responses of Two Different BFR Training Protocols Using Either an Autoregulated Pressure or a Non-autoregulated Pressure
Brief Title: Perceptual, Hemodynamic and Cardiovascular Responses of Two Different BFR Training Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BC-11035
Record Dates: First submitted 2021-11-09; First posted 2021-12-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Blood Flow Restriction; Strength training; Cardiovascular safety; Hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Autoregulated cuff (Experimental): two sessions in which an autoregulated cuff will be used to adapt the pressure in order to keep the total pressure given constant. First session will be within a 30-15-15-15 reps protocol, the second session will be performed until max fatigue.
  Interventions: Device: Autoregulated Blood Flow Restriction Cuff (smart-cuff pro devices, acting as pressurized tourniquet) combined with low load strength training
- non-autoregulated cuff (Active Comparator): two sessions in which an non-autoregulated cuff will be used. In these two sessions, the pressure will not be adapted. Consequently, during each muscle contraction the pressure will rise because the cuff is not autoregulated. First session will be within a 30-15-15-15 reps protocol, the second session will be performed until max fatigue.
  Interventions: Device: Non-autoregulated blood flow restriction cuff ((smart-cuff pro devices, acting as pressurized tourniquet) combined with low load strength training)

INTERVENTIONS:
Device: Autoregulated Blood Flow Restriction Cuff (smart-cuff pro devices, acting as pressurized tourniquet) combined with low load strength training — This group will undergo 2 sessions consisting of a low load leg extension exercise combined with a pressurized tourniquet which autoregulates so when the quadriceps muscle contracts, the total amount of pressure doesn't increase, as the tourniquet will lower the pressure to keep the total amount of pressure constant.
  Other Names: Kaatsu; Partial vascular occlusion
  Arms: Autoregulated cuff
Device: Non-autoregulated blood flow restriction cuff ((smart-cuff pro devices, acting as pressurized tourniquet) combined with low load strength training) — This group will undergo 2 sessions consisting of a low load leg extension exercise combined with a pressurized tourniquet which does not autoregulate so when the quadriceps muscle contracts, the total amount of pressure will increase, as the tourniquet will not lower the pressure to keep the total amount of pressure constant.
  Other Names: Kaatsu; Partial vascular occlusion
  Arms: non-autoregulated cuff

SUMMARY:
BFR training is growing in popularity and a variety of devices are on the market for clinical use. One way in which it is thought that BFR resistance training safety can be increased is by using a BFR cuff that regulates the applied pressure to the limb during each repetition. This is thought to reduce perceptual, hemodynamic and cardiovascular responses to non-autoregulated approaches, theoretically increasing long-term compliance and safety with BFR training.

DETAILED DESCRIPTION:
BFR training is growing in popularity and a variety of devices are on the market for clinical use. One way in which it is thought that BFR resistance training safety can be increased is by using a BFR cuff that regulates the applied pressure to the limb during each repetition. This is thought to reduce perceptual, hemodynamic and cardiovascular responses to non-autoregulated approaches, theoretically increasing long-term compliance and safety with BFR training.

However, only one study has directly compared the effect of an autoregulated vs. non-autoregulated and their design did not standardize the cuff width between the autoregulated and the non-autoregulated cuff, potentially leading to differences in observed outcomes. That study concluded that autoregulated cuffs better manage the hemodynamic and perceptual responses to non-failure training protocols while providing a more accurate cuff-limb interface pressure, thus increasing safety profile. Moreover, BFR resistance training is commonly performed to failure so it is unknown whether the use of regulated pressures influences fatiguability or alters perceptual, cardiovascular and hemodynamic responses compared to a non-autoregulated cuff.

Therefore, the purpose of this study is to compare the perceptual, hemodynamic and cardiovascular responses using either an autoregulated pressure or a non-autoregulated pressure during a 20% 1RM leg extension non-failure and failure protocol in healthy, recreationally active male and female participants (without any history of BFR training) using the SmartTools Pro model (a device able to be autoregulated and non-autoregulated based on setting, providing an ability to directly compare autoregulation to non-autoregulation with a cuff of similar width).

Each participant will perform one familiarization session to determine 1RM, take baseline data for participant characteristics including limb occlusion pressure and relevant hemodynamic and cardiovascular measures, acclimate to the non-failure protocol without blood flow restriction and anchor perceptual baselines. Following familiarization session and at least 6 days between sessions, the dominant leg of each participant will be randomized to either the autoregulated or non-autoregulated pressure setting. Each participant will perform 4 sets of exercise applied in a continuous application setting using a commonly recommended protocol of 30-15-15-15 using a 2 second concentric/2 second eccentric tempo with 30-45 seconds of interset rest. The BFR cuff will either be set to autoregulation or non-autoregulated pressure setting. Following completion of the protocol, with the cuffs still inflated, all variables will be assessed again before deflating. Participants will return to the lab at least 6 days later at a similar time and perform the same protocol with the opposite condition.

To assess the differences in all relevant outcome measures during a failure routine, the same protocol will be completed 6 days later with each participant randomized to either the autoregulated or non-autoregulated group. Participants will complete a similar resistance training program using 4 sets to volitional fatigue instead of the non-failure protocol. The data provided within this study could greatly inform clinical practice if responses to non-autoregulated cuff applications in both non-failure and failure routines are heightened compared to autoregulated cuff applications. This study will also provide preliminary data for application in clinical populations such as those with knee osteoarthritis as well as applying a similar strategy to healthy populations in the upper extremity to determine if similar responses exist between limbs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Be motivated to visit Ghent University Hospital 5 times for 30 minutes

Exclusion Criteria:

* Suffering from a neuromuscular disease, affecting lower limbs
* Reduced functioning or pain in the dominant leg
* Taking pain medication
* Previous cardiovascular surgery affecting lower limbs
* Symptomatic cardiovascular or hemodynamic suffering
* Pregnant
* Increased risk for DVT (genetic or history of)
* Not being able to perform physical activities, for whatever (medical) reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
Change in heart rate | 5 weeks
  Effect of leg extension exercise with blood flow restriction on the cardiovascular system
Change in blood pressure | 5 weeks
  Effect of leg extension exercise with blood flow restriction on the hemodynamic system
Change in rate of perceived exertion (RPE) | 5 weeks
  What is the perception of the patient when doing leg extensions with BFR

SECONDARY OUTCOMES:
Change in 1 repetition maximum | 5 weeks
  heighest weight a participant can lift by doing a leg extension
Change in fatiguability | 5 weeks
  What is the amount of weight a participant can lift during a whole session.
change in delayed onset muscle soreness | 5 weeks
  Does the participant feels stiff/sore 24 hours after the exercise

CONTACTS AND LOCATIONS:
Overall Officials: Erik Witvrouw, Prof. dr., Study Chair — University Ghent
Locations (1):
- University Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request.
Supporting Information: Study Protocol, ICF